CLINICAL TRIAL: NCT04650568
Title: A Prospective Randomized Trial of Biologic Augmentation With Mesenchymal Stem Cells in Patients Undergoing Anterior Cruciate Ligament Reconstruction
Brief Title: Biologic Augmentation With Mesenchymal Stem Cells in Patients Undergoing Anterior Cruciate Ligament Reconstruction
Acronym: BMAC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17082504
Record Dates: First submitted 2017-12-04; First posted 2020-12-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Rupture
Keywords: Anterior Cruciate Ligament; ACL; Stem Cell; Mesenchymal stem cells; biologic; augmentation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient remains blinded throughout trial. Imaging evaluator will be blinded to which study arm the patient belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mesenchymal Stem Cell Recipient (Experimental): Patients in this group will receive between 1-4 ml of bone marrow aspirate concentrate (BMAC) containing mesenchymal stem cells (MSCs) obtained from their iliac crest. A small incision will be made on the anterior superior iliac spine in order to withdraw the aspirate. The aspirate will be ran through a centrifuge in order to isolate the BMAC containing MSCs. The BMAC will be injected into the ACL allograft prior to implanting into the patient.
  Interventions: Device: Autologous Bone Marrow Derived Mesenchymal Stem Cells
- Control Sham Incision (Placebo Comparator): Patients will receive a sham incision on the anterior superior iliac spine where the bone marrow aspirate is obtained in the the experimental group. This ensures proper blinding. The patient will receive the normal standard of care.
  Interventions: Other: Sham incision

INTERVENTIONS:
Device: Autologous Bone Marrow Derived Mesenchymal Stem Cells — Autologous Bone Marrow Derived Mesenchymal Stem Cells injected into the ACL allograft prior to graft implantation.
  Other Names: Sham Incision
  Arms: Mesenchymal Stem Cell Recipient
Other: Sham incision — Small incision over the site where bone marrow aspirate would have been obtained
  Arms: Control Sham Incision

SUMMARY:
This study will evaluate the efficacy of biologic augmentation of ACL reconstruction with bone marrow derived mesenchymal stem cells as measured by magnetic resonance imaging to detect graft healing and integration. Secondary endpoints will include validated patient reported outcome measures, as well as functional outcome using objective examination findings.

DETAILED DESCRIPTION:
Introduction

Anterior cruciate ligament (ACL) tears are a common and devastating injury among young athletes, and re-injury poses significant threats to both successful return to play and long term outcomes. Graft healing during ACL reconstruction (ACLR) is a slow biologic process, that involves graft incorporation into bone tunnel sites, as well as intra-articular graft remodeling . The intra-articular graft remodeling process is known as ligamentization, and occurs in three phases after ACLR. The first phase of early healing occurs between 0 and three months, the second phase occurs between 6 months and one year, and the final phase of maturation occurs after 1 year when the graft appears very similar to the native ACL. The studies that defined these time points biopsied human bone-patella tendon-bone (BTB) ACL autografts at different postoperative points, and described changes occurring over time in regards to vascularization, cellular aspects, and appearance of the extracellular matrix in comparison to control ACLs . Unlike animal models which display a necrotic stage, grafts in human models undergo an early vascular invasion, associated with fibroblasts that are converted to a hyper-cellular matrix with only focalized areas of necrosis . This process occurs as early as 3 weeks postoperatively, and increases over time as areas similar to the native patellar tendon with mature collagen and metabolically quiescent cells decrease . This process is the limiting factor in graft healing for bone-patella tendon-bone (BTB) grafts, as osteointegration occurs earlier .

The processes of osteointegration and ligamentization are responses to the new intrasynovial milieu and physical forces that the new graft is exposed to. During these healing and restructuring processes, failure load and stiffness of grafts decreases by up to 24% at 7 weeks, before strengthening to their potential . This contributes to the long recovery period for ACLR, and the risk of re-rupture during this period. Advances in biologic adjuncts to accelerate and improve this healing process would have a significant impact on the management of ACL injuries.

Recently, biologic preparations of various growth factors have been developed to safely and effectively treat a variety of musculoskeletal conditions, including tendinopathies and arthritis . Bone marrow aspirate concentrate (BMAC) consists of undifferentiated mesenchymal stem cells that are concentrated and applied to the injury site . Previous studies have demonstrated this treatment to offer the pluripotent potential of the cells to impact healing, regeneration, biomechanical strength, and reducing bone-tunnel enlargement . Investigators have demonstrated that mesenchymal stem cell reinforced grafts had a significantly higher failure load and stiffness as early as 8 week post-operation in a rabbit model, suggesting an added benefit of advanced healing . Using BMSCs can offer a novel method to enhance tendon graft osteointegration. While there have been numerous laboratory studies researching the effect of mesenchymal stem cells, there lacks evidence in translation to the clinical setting. Silva et al performed a study where they injected bone marrow derived stem cells (BMSCs) into patellar tendon grafts to examine for increased graft-to-bone tunnel integration. They did not find a significant difference of tunnel integration on MRI imaging, but they did not examine the intra-articular portions for the effect on the ligamentization process, nor did they examine the effect on clinical examination and patient reported outcomes .

Quantitative MRI is a non-invasive method to interrogate tissue properties and evaluate the biochemical composition of tissues. The T2* sequence gives information regarding tissue graft volume, water content, fiber alignment, and tissue density. Median grayscale values (a measure to determine tissue quality)can also be correlated to maximum failure load, yield load, and linear stiffness of grafts in a porcine model. Increases in MRI signals in ACL grafts have been found to be time dependent, becoming well established by three months, particularly at the distal intra-articular portion near the tibial tunnel . These changes have not been shown previously to be predictive of graft failure, but Investigators have recently also confirmed that normalized T2* signal intensity values of ACL grafts have significant correlation with knee instability related to ligamentization and tunnel healing.

A recent study examined intra-articular graft maturation after platelet-rich plasma gel (PRPG) application, with MRI at month intervals from 3-12 months postoperatively. The intra-articular segment was divided in a proximal, middle, and distal segment, on a scale from 0-3 ranging from completely homogenous to severely heterogeneous. The mean time to obtain completely homogenous bone-patella tendon-bone (BTB) graft was 109 days for the PRPG group, and 363 for the control group 8.

We propose using quantitative magnetic resonance (MR) imaging with T2* mapping to investigate if BMAC treatment at time of ACL reconstruction can accelerate the graft maturation and healing process. We will perform a randomized controlled trial of patients undergoing ACL reconstruction with bone-patellar tendon-bone allograft evaluating the T2* weighted MRI changes of the graft at 3 and 9 months after surgical reconstruction. Additionally, we will obtain patient-reported outcome measures from this cohort to evaluate if BMAC treatment imparts a clinically-significant effect on ACL reconstruction.

Study Rationale

This study will evaluate the efficacy of biologic augmentation of ACL reconstruction with BMSCs as measured by magnetic resonance imaging to detect graft healing and integration. Secondary endpoints will include validated patient reported outcome measures, as well as functional outcome using objective examination findings.

Hypothesis

The hypotheses of this study are that there will be improved graft healing and integration at three and nine months as measured by decreased signal intensity and heterogeneity on T2* MRI following administration of BMAC during ACL reconstruction compared to the control group. Additionally, patient reported outcomes and physical examination findings will be significantly improved at an earlier time in those who receive the BMAC treatment to their allograft compared to the control group.

Study Plan

This study will be a prospective randomized trial of patients undergoing arthroscopic reconstruction of full thickness anterior cruciate ligament (ACL) tears. All patients who sign consent and undergo full thickness ACL reconstruction will be enrolled in the study. Enrollment will continue until 32 patients, 16 in each group, are enrolled. Follow-up will take place at 6 weeks, 3 months, 6 months, 9 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* 18-60 years of age with acute ACL injury (<6 months from time of injury to reconstruction) and undergoing reconstruction with patellar tendon allograft
* Written informed consent is obtained

Exclusion Criteria:

* Revision Surgery
* Prior history of knee surgery
* Concomitant ligamentous injury
* Inability to obtain an MRI
* Inability to participate in follow-up for the study
* Any patient lacking decisional capability
* Diagnosed musculoskeletal cancer or any diagnosed cancer, other than
* musculoskeletal if not on long term remission (e.g. at least 5 years or negative biopsy at last exam), except basal cell carcinoma
* Patients who are at higher risk for post-surgical bleeding (e.g., bleeding disorder taking anticoagulants except low dose aspirin) or post-surgical infection (e.g., taking immunosuppressants; have a severe infection or a history of serious infection or use of systemic steroids)
* Known history of HIV, or has active Hepatitis B or active Hepatitis C
* Alcohol and drug (medication) abuse
* Pregnant or breast feeding women. Pregnancy as determined by a positive pregnancy test prior to procedure. Females of childbearing potential must agree to use an acceptable birth control method during study participation.
* Patients that have received PRP, other platelet-based product, or investigational treatment in another cell/biologic study for the target knee in the 12 months prior to the injection procedure
* Any clinically significant finding that would place the patient at health risk, impact the study, or affect the completion of the study
* Any psychiatric illness that would prevent comprehension of the details and nature of the study and interfere with follow-up clinic visits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Signal to Noise Quotient | 9 months
  Signal intensity of the ACL graft on T2 weighted MRI imaging compared to a reference structures' signal intensity

SECONDARY OUTCOMES:
Side to side difference in anterior tibial translation | 6 weeks, 3 months, 6 months, 9 months, 1 year
  Anterior tibial translation measured by (Knee laxity Testing device) KT-1000 Arthrometer
Patient reported outcomes- Tegner Score | 3 months, 6 months, 9 months, 12 months, 24 months
  Patient reported outcome measure for patients receiving arthroscopic knee surgery
Patient reported outcomes- Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr) | 3 months, 6 months, 9 months, 12 months, 24 months
  Patient reported outcome measure for patients receiving arthroscopic knee surgery
Patient reported outcomes- International Knee Documentation Committee (IKDC) Score | 3 months, 6 months, 9 months, 12 months, 24 months
  Patient reported outcome measure for patients receiving arthroscopic knee surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No